CLINICAL TRIAL: NCT00765128
Title: The Efficacy of Continuous Intravenous Ketorolac for Postoperative Pain in Percutaneous Nephrolithotomy: a Double Blinded Randomized Placebo Controlled Trial
Brief Title: Intravenous Ketorolac for Postoperative Pain in Percutaneous Nephrolithotomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Mitchell R. Humphreys, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-000747 PNL
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Results first posted 2012-01-27 (Estimated); Last update posted 2012-01-27 (Estimated); Status verified 2011-12

CONDITIONS: Renal Calculus; Kidney Stones
Keywords: Percutaneous; Nephrolithotomy; Kidney stones
MeSH Terms: conditions — Kidney Calculi | interventions — Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketorolac (Experimental): 90 mg ketorolac in 1 L of normal saline infused at 40-120 mL/hr for 18.5-23 hours beginning 0.5 hours after the end of surgery.
  Interventions: Drug: Ketorolac
- Placebo (Placebo Comparator): 1 L of normal saline infused at 40-120 mL/hr for 18.5-23 hours beginning 0.5 hours after the end of surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketorolac — 90 mg ketorolac in 1 L of normal saline infused at 40-120 mL/hr for 18.5-23 hours beginning 0.5 hours after the end of surgery.
  Other Names: Toradol; Acular
  Arms: Ketorolac
Drug: Placebo — 1 L of normal saline infused at 40-120 mL/hr for 18.5-23 hours beginning 0.5 hours after the end of surgery.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether continuous intravenous ketorolac infusion reduces pain in patients who are having percutaneous nephrolithotomy for kidney stone disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing percutaneous nephrolithotomy for kidney stone disease

Exclusion Criteria:

* History of nonsteroidal antiinflammatory drug allergy
* Asthma
* History of long-term opioid use
* Intraoperative blood loss greater than 300 mL
* Postoperative hemodynamic instability
* Active peptic ulcer disease
* Advanced renal impairment (Creatinine > 2.0 mg/dL)
* Bleeding diathesis
* Current use of probenecid
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell R. Humphreys, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Grimsby GM, Andrews PE, Castle EP, Nunez R, Mihalik LA, Chang YH, Humphreys MR. Long-term renal function after donor nephrectomy: secondary follow-up analysis of the randomized trial of ketorolac vs placebo. Urology. 2014 Jul;84(1):78-81. doi: 10.1016/j.urology.2014.04.009. PMID 24976224
- [Derived] Grimsby GM, Conley SP, Trentman TL, Castle EP, Andrews PE, Mihalik LA, Hentz JG, Humphreys MR. A double-blind randomized controlled trial of continuous intravenous Ketorolac vs placebo for adjuvant pain control after renal surgery. Mayo Clin Proc. 2012 Nov;87(11):1089-97. doi: 10.1016/j.mayocp.2012.07.018. Epub 2012 Oct 8. PMID 23058854

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from October 2008 to November 2010.
Period: Overall Study
Arm/Group | Ketorolac | Placebo
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketorolac | Placebo | Total
Number analyzed (Participants) | 8 | 9 | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 59.0 (8.0) | 62.0 (9.8) | 60.6 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Pain 'Right Now'
Description: Visual analog scale score for pain on a scale from 0 = None to 10 = Worst.
Time Frame: 24 hours after the end of surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac | Placebo
Number analyzed (Participants) | 8 | 9
units on a scale | 1.0 (1.2) | 0.9 (1.5)

2. Primary Outcome: Morphine Equivalents of Concomitant Pain Medication
Description: The morphine equivalent is a unit of measure to compare the efficacy of different types of opioids (narcotics). The patients were allowed to take additional pain medication in addition to either study drug or placebo. This outcome measure reports the amount of morphine (in mg) equivalent to the amount of concomitant pain medication used by the patient.
Time Frame: 24 hours after the end of surgery
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Ketorolac | Placebo
Number analyzed (Participants) | 8 | 9
mg | 15 (33) | 10 (14)

ADVERSE EVENTS:
Time Frame: Adverse events were noted during hospitalization (approximately 4 days).
Arm/Group | Ketorolac | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 8/8 | 8/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketorolac (N=8) | Placebo (N=9)
Anaemia (Blood and lymphatic system disorders) | 7 (7) | 2 (2)
Hypochloraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Blood Urea Nitrogen Increased (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Nonprotein Nitrogen Increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Leucopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Monocytopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Hyperchloraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Lymphadenopathy Cervical (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Granulocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypocapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes